CLINICAL TRIAL: NCT07240168
Title: Drug Retention in Vedolizumab-treated Patients With Active UC After the Addition of Adjunct CurQD: A Retrospective Cohort Study
Brief Title: CurQD as Add-On Therapy in Vedolizumab-Treated Ulcerative Colitis Patients: Retrospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Evinature Ltd. (Other)
Collaborators: Sheba Medical Center (Other Government); Takeda Pharmaceuticals U.S.A., Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIR-2024-200598
Record Dates: First submitted 2025-09-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Curcumin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1 (VDZ + CurQD): Patients with ulcerative colitis on Vedolizumab who initiated CurQD as adjunct therapy.
  Interventions: Dietary Supplement: CurQD (Curcumin + QingDai combination)

INTERVENTIONS:
Dietary Supplement: CurQD (Curcumin + QingDai combination) — Patients received CurQD in addition to Vedolizumab

SUMMARY:
This study aims to evaluate whether adding CurQD, a nutraceutical composed of Curcumin and QingDai, improves treatment outcomes in patients with active ulcerative colitis (UC) who are already receiving Vedolizumab but still have ongoing disease activity. The study will use de-identified patient records collected through Evinature's global data platform. We will examine whether the addition of CurQD helps patients stay on Vedolizumab longer, improves symptoms and biomarkers, and increases satisfaction with treatment.

DETAILED DESCRIPTION:
Curcumin and QingDai, (Indigo, QD) are two herbal traditional medicine compounds which have been investigated for their use in mild-moderate and moderate-severe UC, respectively. A combination of Curcumin and QD (CurQD), which was developed at Sheba Medical Center to maximize clinical efficacy while reducing long-term high-dose QD exposure, has been used in clinical practice in Israel since 2015 and has gained wide acceptance by UC patients and IBD experts [1,2]. In two multi-center retrospective studies, CurQD was found effective in inducing clinical and biomarker remission in both adult and pediatric patients, including in patients who were refractory to biologic and/or small molecules [3,4], and recent evidence from a pediatric cohort in the U.S also documented intestinal sonographic response to CurQD [5]. In a placebo-controlled randomized trial from Israel and Greece, CurQD was found superior to placebo in inducing and maintaining clinical and endoscopic remission without any safety signals [6,7]. Moreover, the study also showed the active compounds in CurQD exerts agonistic up-regulation of Aryl-hydrocarbon Receptor pathway in the rectal mucosa [6], supporting its unique non-immunosuppressive mode-of-action. Subsequently, CurQD has been increasingly used by IBD experts in academic centers in the USA and elsewhere as Add-on therapy in patients with partial or non-response to biologics and/or small molecules medications. Recently, CurQD became the first and only nutraceutical to date to pass the CCFA Ingestible committee examination of supporting clinical and scientific data to allow its endorsement by the CCFA. Collectively, these data provide the rationale for exploring large scale population-based impact of combining CurQD with a biologic.

The present retrospective cohort study will interrogate the Evinature GDPR HIPAA compliant database to identify patients who started CurQD while being treated with VDZ. The study will investigate the clinical benefit of adding CurQD in combination with VDZ, in patients partially responding or not-responding to VDZ.

ELIGIBILITY:
Inclusion Criteria:

* Age >8 years
* Diagnosis of ulcerative colitis (self-reported)
* Completed Evinature clinical assessment between April 1, 2022, and cutoff date
* Vedolizumab treatment at baseline
* Active disease at entry (SCCAI ≥3 or PRO-2 ≥2 with RB ≥1)
* Initiated CurQD at entry

Exclusion Criteria:

* Vedolizumab for indications other than UC
* Unclear medication status at baseline
* Not active disease when starting CurQD

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise adult and pediatric (age > 8 years-old) UC patients with active disease while on VDZ treatment who start CurQD combo therapy concomitantly with VDZ
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Retaining Vedolizumab Treatment at Week 12 Following Addition of CurQD | Week 12
  Count of participants who remain on vedolizumab (VDZ) at Week 12 after initiating adjunct CurQD. Baseline clinical activity is defined as SCCAI ≥3 or PRO-2 ≥2 with rectal bleeding ≥1. Percentages will also be calculated relative to the number of participants with Week 12 data.

SECONDARY OUTCOMES:
Number of Participants Retaining Vedolizumab at Week 30 | Week 30
  Count of participants with ≥30 weeks of follow-up who remain on VDZ at Week 30 after starting CurQD. Percentages will also be calculated relative to the number of participants with Week 30 data.
Number of Participants Retaining Vedolizumab at Week 54 | Week 54
  Count of participants with ≥54 weeks of follow-up who remain on VDZ at Week 54 after starting CurQD. Percentages will also be calculated relative to the number of participants with Week 54 data
Number of Participants Achieving Clinical Remission at Week 12 | Week 12
  Clinical response is defined as SCCAI decrease ≥3, or PRO-2 decrease ≥2 with RB = 0 and SF ≤1, among participants with available baseline and follow-up values. Percentages will also be calculated relative to the number of participants with Week 12 clinical data.
Number of Participants Achieving Clinical Response at Week 54 | Week 54
  Same response definition as above. Percentages will also be calculated relative to the number of participants with Week 54 clinical data.
Number of Participants in Clinical Remission at Week 12 | Week 12
  Clinical remission defined as SCCAI ≤2 or PRO-2 = 0. Percentages will also be calculated relative to the number of participants with Week 12 clinical data.
Number of Participants in Clinical Remission at Week 54 | Week 54
  Same remission definition as above. Percentages will also be calculated relative to the number of participants with Week 54 clinical data.
Number of Participants Reporting Satisfaction with CurQD + Vedolizumab (VAS 1-10) | Week 12
  Number of participants providing a satisfaction score using a 1-10 Visual Analog Scale (VAS) after using CurQD + VDZ. Percentages will also be calculated relative to the number of participants who completed the VAS assessment.
Number of Participants Achieving Fecal Calprotectin (FCP) Response | Up to Week 54
  FCP response defined as ≥50% reduction from baseline among participants with baseline FCP ≥250 mcg/g and available follow-up FCP. Percentages will also be calculated relative to the number of participants with FCP measurements.
Number of Participants Achieving Fecal Calprotectin (FCP) Remission | Up to Week 54
  FCP remission defined as FCP <150 mcg/g among participants with baseline FCP ≥250 mcg/g, following STRIDE II and GEMINI-I guidance. Percentages will also be calculated relative to the number of participants with FCP measurements.
Number of Participants Experiencing Treatment-Emergent Adverse Events | Baseline through Week 54
  Number and type of adverse events occurring during combined CurQD + VDZ therapy. Percentages will also be calculated relative to the number of participants exposed to both therapies.
Sensitivity Analysis: Number of Participants Retaining Vedolizumab at Week 12 with Baseline SCCAI ≥6 | Week 12
  Same definition as the primary endpoint but limited to participants with moderate-severe disease (baseline SCCAI ≥6). Percentages will also be calculated relative to the number of participants in this subgroup with Week 12 data.

CONTACTS AND LOCATIONS:
Overall Officials: Shomron Ben-Horin, Study Director — Evinature Ltd.
Locations (1):
- Evinature, Binyamina, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reinisch W, Bressler B, Curtis R, Parikh A, Yang H, Rosario M, Roseth A, Danese S, Feagan B, Sands BE, Ginsburg P, Dassopoulos T, Lewis J, Xu J, Wyant T. Fecal Calprotectin Responses Following Induction Therapy With Vedolizumab in Moderate to Severe Ulcerative Colitis: A Post Hoc Analysis of GEMINI 1. Inflamm Bowel Dis. 2019 Mar 14;25(4):803-810. doi: 10.1093/ibd/izy304. PMID 30295811
- [Result] Turner D, Ricciuto A, Lewis A, D'Amico F, Dhaliwal J, Griffiths AM, Bettenworth D, Sandborn WJ, Sands BE, Reinisch W, Scholmerich J, Bemelman W, Danese S, Mary JY, Rubin D, Colombel JF, Peyrin-Biroulet L, Dotan I, Abreu MT, Dignass A; International Organization for the Study of IBD. STRIDE-II: An Update on the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) Initiative of the International Organization for the Study of IBD (IOIBD): Determining Therapeutic Goals for Treat-to-Target strategies in IBD. Gastroenterology. 2021 Apr;160(5):1570-1583. doi: 10.1053/j.gastro.2020.12.031. Epub 2021 Feb 19. PMID 33359090
- [Result] Abreu MT, Rowbotham DS, Danese S, Sandborn WJ, Miao Y, Zhang H, Tikhonov I, Panaccione R, Hisamatsu T, Scherl EJ, Leong RW, Arasaradnam RP, Afif W, Peyrin-Biroulet L, Sands BE, Marano C. Efficacy and Safety of Maintenance Ustekinumab for Ulcerative Colitis Through 3 Years: UNIFI Long-term Extension. J Crohns Colitis. 2022 Aug 30;16(8):1222-1234. doi: 10.1093/ecco-jcc/jjac030. PMID 35239968
- [Result] Walsh AJ, Ghosh A, Brain AO, Buchel O, Burger D, Thomas S, White L, Collins GS, Keshav S, Travis SP. Comparing disease activity indices in ulcerative colitis. J Crohns Colitis. 2014 Apr;8(4):318-25. doi: 10.1016/j.crohns.2013.09.010. Epub 2013 Oct 10. PMID 24120021
- [Result] Ben-Horin S, Salomon N, Yanai H, Kopylov U. Letter: Change in Bowel Urgency in Active Ulcerative Colitis Patients Treated with Curcumin-QingDai (CurQD): A Post Hoc Analysis of a Randomized Placebo-Controlled Trial. J Crohns Colitis. 2025 Mar 5;19(3):jjae147. doi: 10.1093/ecco-jcc/jjae147. No abstract available. PMID 39279191
- [Result] Ben-Horin S, Salomon N, Karampekos G, Viazis N, Lahat A, Ungar B, Eliakim R, Kuperstein R, Kriger-Sharabi O, Reiss-Mintz H, Yanai H, Dotan I, Zittan E, Maharshak N, Hirsch A, Weitman M, Mantzaris GJ, Kopylov U. Curcumin-QingDai Combination for Patients With Active Ulcerative Colitis: A Randomized, Double-Blinded, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2024 Feb;22(2):347-356.e6. doi: 10.1016/j.cgh.2023.05.023. Epub 2023 Jun 9. PMID 37302449
- [Result] Chavannes M, Kandavel P, Danialifar T, Dillman J, Polk DB, Clinical, biochemical and intestinal ultrasonography response to curcumin-QIngDai (CurQD) combination in pediatric patients with inflammatory bowel disease: A case series, Inflam Bowel Dis 2024; 30, Suppl 1, Pages S18-S19, https://doi.org/10.1093/ibd/izae020.044
- [Result] Nachum NL, Salomon N, Yerushalmy-Feler A, Weintraub Y, Yogev D, Granot M, Haberman Y, Ben-Horin S, Weiss B. The efficacy of curcumin/Qing Dai combination in children with active ulcerative colitis: a multicenter retrospective cohort study. Front Pediatr. 2024 Sep 27;12:1342656. doi: 10.3389/fped.2024.1342656. eCollection 2024. PMID 39403348
- [Result] Yanai H, Salomon N, Lahat A, Ungar B, Eliakim R, Kriger-Sharabi O, Reiss-Mintz H, Koslowsky B, Shitrit AB, Tamir-Degabli N, Dotan I, Zittan E, Maharshak N, Hirsch A, Ben-Horin S, Kopylov U. Real-world experience with Curcumin-QingDai combination for patients with active ulcerative colitis: A retrospective multicentre cohort study. Aliment Pharmacol Ther. 2023 Jul;58(2):175-181. doi: 10.1111/apt.17538. Epub 2023 May 8. PMID 37157131
- [Result] Zittan E, Mahajna H, Salomon N. Attitudes Toward Integrative Medicine in Inflammatory Bowel Disease: A Survey Among Israeli Inflammatory Bowel Disease Experts. Inflamm Bowel Dis. 2023 Sep 1;29(9):e35-e36. doi: 10.1093/ibd/izad072. No abstract available. PMID 37116868
- [Result] Ben-Horin S, Kopylov U, Salomon N. Curcumin-QingDai Combination as Treatment for Moderate-Severe Ulcerative Colitis. Case Rep Gastroenterol. 2022 Sep 20;16(3):563-568. doi: 10.1159/000526646. eCollection 2022 Sep-Dec. PMID 36824698